CLINICAL TRIAL: NCT05437809
Title: Biobehavioral Reward Responses Associated With Consumption of Nutritionally Diverse Ultra-Processed Foods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Oregon Research Institute Community and Evaluation Services (Unknown)
Responsible Party: Principal Investigator, elafata@ori.org, Research Scientist, Oregon Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: K23DK129825 (NIH)
Record Dates: First submitted 2022-06-19; First posted 2022-06-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overeating; Food Addiction
Keywords: Ultra-processed foods; Food reward
MeSH Terms: conditions — Obesity; Hyperphagia; Food Addiction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UPF high in fat and refined carbohydrates (Other): This test snack condition consists of ultra-processed foods high in both fat and refined carbohydrates.
  Interventions: Other: Intake of nutritionally diverse ultra-processed foods
- UPF high in fat (Other): This test snack condition consists of ultra-processed foods high in fat.
  Interventions: Other: Intake of nutritionally diverse ultra-processed foods
- UPF high in refined carbohydrates (Other): This test snack condition consists of ultra-processed foods high in refined carbohydrates.
  Interventions: Other: Intake of nutritionally diverse ultra-processed foods
- MPF high in fat or carbohydrates (Other): This test snack condition consists of minimally processed foods naturally high in either fat or carbohydrates.
  Interventions: Other: Intake of nutritionally diverse ultra-processed foods

INTERVENTIONS:
Other: Intake of nutritionally diverse ultra-processed foods — All participants will attend four food consumption assessment visits where, at each visit, they will be asked to consume a standardized snack portion of: 1) ultra-processed foods (UPFs) high in both fat and refined carbohydrates (UPF+FRC), 2) UPF high in fat (UPF+F), 3) UPF high in refined carbohydrates (white flour, sugar) (UPF+RC), or 4) minimally processed foods. The order of the four food consumption assessment visits will be randomized and counterbalanced across participants, who will each consume all the test snacks across the four appointments.

SUMMARY:
The changing food environment, with increasingly abundant ultra-processed food (UPF) options, may directly contribute to rising rates of obesity, though it is unknown which ingredients in UPF elevate their reinforcing nature in a way that may lead to overconsumption. The proposed study is the first to systematically examine differences in the rewarding characteristics of and physiological and metabolic responses to UPFs that are high in fat, refined carbohydrates (like sugar), or both. Understanding the biobehavioral underpinnings that enhance the reinforcing potential of ingredients in UPF (e.g., fat vs. refined carbohydrates) can inform novel intervention targets for the treatment of overeating and obesity.

DETAILED DESCRIPTION:
The abundance of ultra-processed foods (UPFs) in our environment has led to excessive calorie intake and been cited as perpetuating the obesity epidemic. UPFs do not exist in nature and are created to maximize palatability through the additions of fat, refined carbohydrates (RC), and/or sodium (e.g., chocolate, potato chips). Emerging research suggests UPFs may be reinforcing akin to rewarding substances like alcohol. However, empirical investigation of which ingredients in UPFs directly motivate overeating is in its nascent stages. This study will be the first to combine biological and behavioral methods used in addiction research with assessments of food reward, to delineate the mechanisms by which fat and RC drive UPF reinforcement and influence future consumption.

Individuals (n=50) with obesity will be recruited for the current study. Participants will attend four appointments (order randomized/counterbalanced) and will consume a snack consisting of 1) UPF high in fat + RC (UPF+FRC), 2) UPF high in fat (UPF+F), 3) UPF high in RC (UPF+RC), or 4) minimally processed foods (MPF). At each assessment, subjective experiences and metabolic responses will be assessed before and up to 120 minutes after consumption of each snack. An ad-libitum eating period for each food condition will follow to evaluate associations of metabolic/behavioral responses with subsequent intake. For five days after each appointment, participants will use ecological momentary assessment (EMA) to assess subjective experiences and real-world reported consumption of UPF+FRC, UPF+F, UPF+RC, and MPF.

ELIGIBILITY:
Inclusion Criteria Men and women Age 18-65 years BMI ≥ 30 kg/m2 Endorse liking the foods included in the compulsory test snacks at a 6 on a scale from 1-10 No history of severe psychiatric illness; current mild to moderate severity of depression, anxiety, or binge eating disorder, determined by the behavioral evaluation and the screening measures will be included Live in the greater Springfield, Oregon area and are willing/able to participate in six in-person assessments Can access and are willing/able to use a smartphone

Exclusion Criteria Medical condition that may limit consumption of compulsory test snack foods or impact metabolic responses to food consumption Type I or II diabetes (HbA1c > 6.5 based on blood test) Uncontrolled hypertension (blood pressure ≥ 140/90 mm Hg) Cardiovascular event (e.g., stroke, myocardial infarction) in the last 12 months Individuals with dietary allergies of aversions to the test snack foods Individuals taking medications that may influence the metabolic responses of interest (e.g., metformin) Individuals who are actively pursuing weight loss or have lost ≥ 5% of their initial weight in the last 6 months Severe symptoms of mood, anxiety, and any severity of thought disorders Severe binge eating disorder or full criteria bulimia Persons with active substance-use disorders Current, active suicidal ideation, and/or a suicide attempt within the past year History of bariatric surgery Women who are nursing, pregnant, or planning to become pregnant in the next three months Self-report current diagnosis of a transferrable blood condition (including HIV, hepatitis B, hepatitis C, or syphilis) Self-report prior history of being dizzy or anxious during blood draws and/or technician not being able to find a vein.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Subjective reward responses to food intake (in lab) | 10 minutes before intake of test snack, during, and 30-, 60-, 90-, and 120 minutes after intake of the test snack.
  Indicators of subjective reward (craving, palatability, hedonic hunger, and mood) will be assessed by participants' self-reports before, during, and after consumption of the test snack at each of the four food consumption appointments. Each facet of subjective reward will be assessed by 100-point visual analog scales ranging from 0-100.
Subjective reward responses to food intake (EMA) | EMA surveys administered over 5 days following each food consumption assessment (20 total days of EMA data)
  Indicators of subjective reward (craving, palatability, hedonic hunger, and mood) will be assessed by participants' self-reports in EMA surveys. Each facet of subjective reward will be assessed by 100-point visual analog scales ranging from 0-100.
Ad libitum consumption | 2 hours after test snack intake at each food consumption assessment.
  Total number of calories consumed from the test snack food during a 15-minute eating period. Calories will calculated by measuring bowls containing the test snacks before and after participant consumption on a digital scale accurate to 0.01 grams. The difference in grams will be converted into the calories that the participant ate.
Daily calorie intake (EMA) | EMA surveys administered over 5 days following each food consumption assessment (20 total days of EMA data)
  Calorie intake will be derived from participants' self-reported food consumption in EMA surveys.
Consumption of UPFs and MPFs (EMA) | EMA surveys administered over 5 days following each food consumption assessment (20 total days of EMA data)
  Trained study staff will calculate the percentage of participants' daily calories from the four food categories (UPF+FRC, UPF+F, UPF+RC, MPF) based on participants' self-reported food consumption in EMA surveys.

SECONDARY OUTCOMES:
Changes in heart rate in response to food intake | 10 minutes before intake of test snack, during, and 30-, 60-, 90-, and 120 minutes after intake of the test snack.
  Manually measured by counting the radial pulse for 15 seconds (timed using a digital stopwatch).
Salivation responses to food intake | 10 minutes before intake of test snack, during, and 30-, 60-, 90-, and 120 minutes after intake of the test snack.
  Participants will spit into a plastic cup for 1 minute and the weight of their saliva will be measured in grams using a digital food scale accurate to 0.01 grams.
Magnitude of metabolic responses to food intake | 10 minutes before intake of test snack, during, and 30-, 60-, 90-, and 120 minutes after intake of the test snack.
  Serial blood draws will be conducted before, during, and after test snack consumption. Samples will be assayed for glucose, insulin, ghrelin, and leptin levels.

OTHER OUTCOMES:
Individual risk factors for enhanced ultra-processed food reward | Tasks administered at baseline assessment (prior to any food consumption appointments) or follow-up assessment (at least one week or up to 2 months after the last food consumption appointment)
  Characteristics known to increase one's reward responsiveness to substances like alcohol will be assessed by behavioral tasks and evaluated as predictors of ultra-processed food reward (delay discounting task to assess impulsivity; Stroop task to assess cognitive functioning; relative reinforcing value task to assess reward value of various foods).

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The project will generate multi-modal data from 50 adults with obesity, including repeated measures of subjective reward responses, physiological and metabolic markers (e.g., heart rate, insulin, glucose, ghrelin, leptin), ecological momentary assessment (EMA) reports, and behavioral task performance (e.g., Stroop, delay discounting, relative reinforcing value). Data will include numeric, categorical, and time-series variables collected across six study visits and four EMA sampling periods. All data will be de-identified and stored in structured formats suitable for statistical analysis.
Supporting Information: Study Protocol, ICF
Time Frame: Data associated with a study publication will be made available upon first publication of the findings. Data will be available indefinitely.
Access Criteria: Dr. LaFata (PI) will be responsible for overseeing the data management and sharing of this project. Dr. LaFata will administer data collection, storage, and repository training to the research coordinator and to any volunteer study staff, who must demonstrate competence in all tasks before commencing their responsibilities. All project staff who use data will have received training in responsible data practices.
  ORI- Community and Evaluation Services will be conducting routine monitoring inspection of randomly selected studies that have indicated a Data and Sharing Management Plan and have received or been awarded funds through NIH and subject to the NIH Data Sharing Policy.